CLINICAL TRIAL: NCT00000543
Title: Oral Calcium in Pregnant Women With Hypertension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Prevention
Other Study IDs: 86; R01HL048846 (NIH)
Record Dates: First submitted 1999-10-27; First posted 1999-10-28 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2002-04

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Hypertension; Pre-Eclampsia; Pregnancy Toxemias; Vascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Hypertension; Pre-Eclampsia; Vascular Diseases | interventions — Dietary Supplements; Calcium

INTERVENTIONS:
Behavioral: dietary supplements
Drug: calcium

SUMMARY:
To determine of providing calcium supplementation to women with pre-existing hypertension reduces the level of blood pressure, requirement for antihypertensive drugs, and incidence of pre-eclampsia.

DETAILED DESCRIPTION:
BACKGROUND:

Maternal and fetal complications are more likely to occur in pregnant women with preexisting hypertension. Alterations in calcium metabolism, the renin angiotensin system, and intracellular free calcium concentration have been identified in this high risk population. The beneficial effects of calcium supplementation on blood pressure and the incidence of superimposed pre-eclampsia may be due to correction of the hormonal and cellular basis for vasoconstriction. The trial sought to prove that oral calcium lowered parathyroid hormone, reduced intracellular free calcium, and decreased vascular endothelin production, resulting in vasodilation and compensatory stimulation of the renin-angiotensin system.

DESIGN NARRATIVE:

Randomized. Double blind. In this observational study, subjects were assigned to two grams of supplemental elemental calcium or to placebo at 13 to 15 weeks gestation. The trial determined the effect of oral calcium supplementation on: the level of blood pressure; the need for antihypertensive drugs; forearm and peripheral vascular resistance; the incidence of maternal complications, including pre-eclampsia and eclampsia; and plasma levels of vitamin D3, ionized calcium, parathyroid, renin activity, angiotensin II, endothelin, nitrate/nitrite, prostacyclins, and intracellular calcium concentrations in lymphocytes and platelets. These variables were measured prior to randomization and every two months throughout pregnancy and the postpartum. Support ended in July 1999.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
Pregnant women with chronic hypertension.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Dates: Start 1993-08; Study Completion 1999-07 (Actual)

REFERENCES:
- [Background] Hojo M, August P. Calcium metabolism in normal and hypertensive pregnancy. Semin Nephrol. 1995 Nov;15(6):504-11. PMID 8588110
- [Background] Hojo M, Suthanthiran M, Helseth G, August P. Lymphocyte intracellular free calcium concentration is increased in preeclampsia. Am J Obstet Gynecol. 1999 May;180(5):1209-14. doi: 10.1016/s0002-9378(99)70618-6. PMID 10329879
- [Background] Curnow KM, Pham T, August P. The L10F mutation of angiotensinogen is rare in pre-eclampsia. J Hypertens. 2000 Feb;18(2):173-8. doi: 10.1097/00004872-200018020-00007. PMID 10694185